CLINICAL TRIAL: NCT06043674
Title: A Phase 2 Study of Glofitamab as Monotherapy or in Combination With Polatuzumab Vedotin, Pirtobrutinib, or Atezolizumab in Richter's Transformation
Brief Title: Phase 2 Study of Glofitamab Monotherapy & With Polatuzumab Vedotin, Pirtobrutinib, or Atezolizumab in Richter's Transformation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christine Ryan (Other)
Collaborators: Genentech, Inc. (Industry); Loxo Oncology, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Christine Ryan, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-429
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Richter's Transformation
Keywords: Chronic Lymphocytic Leukemia; CLL; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — glofitamab; obinutuzumab; polatuzumab vedotin; atezolizumab; tocilizumab; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy Cohort: Obinutuzumab and Glofitamab (Active Comparator): Study procedures will be conducted as follows:
  * Baseline visit with screening procedures, including bone marrow biopsy and Positron Emission Tomography (PET) or Computed Topography (CT) scans.
  * PET/CT scans after 4, 8, and 12 cycles of therapy and at 6 and 15 months after end-of-treatment.
  * Cycle 1:
    * Day 1, 2, and 7 of 21- day Cycle: Predetermined dose of Obinutuzumab 1x daily.
    * Day 8 and 15 of 21- day Cycle: Predetermined dose of Glofitamab 1x daily. Hospitalization will be required for initial dose and post-dose observation.
  * Cycle 2 - 12
    --Day 1 of 21-day Cycle: Predetermined dose of Glofitamab 1x daily. Hospitalization will be required for second dose and post-dose observation
  * End of treatment visit.
  * Follow up visits: for months 10 - 24, visits will be every 3 months. For months 25 - 60 visits will be every 6 months.
  * After completion of a 10-patient safety lead-in cohort, enrollment will open to the other two cohorts.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab
- Combination A Group: Obinutuzumab, Glofitamab, and Polatuzumab Vedotin (Experimental): Study procedures will be conducted as follows:
  * Baseline visit with screening procedures, including bone marrow biopsy and PET/CT scans.
  * PET/CT scans after 4, 8, and 12 cycles of therapy and at 6 and 15 months after end-of-treatment.
  * Cycle 1:
    * Day 1, 2, and 7 of 21- day Cycle: Predetermined dose of Obinutuzumab 1x daily.
    * Day 8 and 15 of 21- day Cycle: Predetermined dose of Glofitamab 1x daily. Hospitalization will be required for initial dose and post-dose observation.
  * Cycle 2 - 7:
    - Day 1 of 21-day Cycle: Predetermined dose of Glofitamab 1x daily. Predetermined dose of Polatuzumab Vedotin 1x daily.
  * Cycle 8 - 12
    - Day 1 of 21-day Cycle: Predetermined dose of Glofitamab 1x daily.
  * End of treatment visit.
  * Follow up visits: for months 10 - 24, visits will be every 3 months. For months 25 - 60 visits will be every 6 months.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Tocilizumab
- Combination B Group: Obinutuzumab, Glofitamab, and Pirtobrutinib (Experimental): Study procedures will be conducted as follows:
  * Baseline visit with screening procedures, including bone marrow biopsy and PET/CT scans.
  * PET/CT scans after 4, 8, and 12 cycles of therapy and at 6 and 15 months after end-of-treatment.
  * Cycle 1:
    * Day 1, 2, and 7 of 21- day Cycle: Predetermined dose of Obinutuzumab 1x daily.
    * Day 8 and 15 of 21- day Cycle: Predetermined dose of Glofitamab 1x daily. Hospitalization will be required for initial dose and post-dose observation.
  * Cycle 2 - 12
    - Day 1 of 21-day Cycle: Predetermined dose of Glofitamab 1x daily. Predetermined dose of Pirtobrutinib 1x daily. Days 2-21 of each cycle: Pirtobrutinib will be taken once daily.
  * End of treatment visit.
  * Follow up visits: for months 10 - 24, visits will be every 3 months. For months 25 - 60 visits will be every 6 months.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab; Drug: Pirtobrutinib
- Combination C Group: Obinutuzumab, Glofitamab, and Atezolizumab (Experimental): Study procedures will be conducted as follows:
  * Baseline visit with screening procedures, including bone marrow biopsy and PET/CT scans.
  * PET/CT scans after 4, 8, and 12 cycles of therapy and at 6 and 15 months after end-of-treatment.
  * Cycle 1:
    * Day 1, 2, and 7 of 21- day Cycle: Predetermined dose of Obinutuzumab 1x daily.
    * Day 8 and 15 of 21- day Cycle: Predetermined dose of Glofitamab 1x daily. Hospitalization will be required for initial dose and post-dose observation.
  * Cycle 2 - 12
    - Day 1 of 21-day Cycle: Predetermined dose of Glofitamab 1x daily. Predetermined dose of Atezolizumab 1x daily.
  * End of treatment visit.
  * Follow up visits: for months 10 - 24, visits will be every 3 months. For months 25 - 60 visits will be every 6 months.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Atezolizumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Glofitamab — "2:1" T-cell bispecific humanized monoclonal antibody, administered via intravenous infusion per protocol.
  Other Names: RO7082859
Drug: Obinutuzumab — Humanized glycoengineered type II anti-CD20 monoclonal antibody, administered via intravenous infusion per protocol.
  Other Names: RO5072759, GA101, GAZYVA, GAZYVARO
Drug: Polatuzumab Vedotin — Antibody-drug conjugate, administered via intravenous infusion per protocol.
  Other Names: Polivy
  Arms: Combination A Group: Obinutuzumab, Glofitamab, and Polatuzumab Vedotin
Drug: Atezolizumab — Humanized immunoglobulin monoclonal antibody, administered via intravenous infusion per protocol.
  Other Names: Tecentriq
  Arms: Combination C Group: Obinutuzumab, Glofitamab, and Atezolizumab
Drug: Tocilizumab — For the treatment of Cytokine Release Syndrome. Recombinant, humanized, anti-human monoclonal antibody, administered via intravenous infusion per protocol.
  Other Names: Actemra
Drug: Pirtobrutinib — Selective inhibitor of BTK, 50 mg or 100 mg tablet, via oral administration per protocol.
  Other Names: Jaypirca
  Arms: Combination B Group: Obinutuzumab, Glofitamab, and Pirtobrutinib

SUMMARY:
This research is being done to evaluate Glofitamab by itself or in combination with Polatuzumab Vedotin, Pirtobrutinib, or Atezolizumab as possible treatments for Chronic Lymphocytic Leukemia (CLL) that has transformed into Richter's Transformation (RT).

The names of the study drugs involved in this research study are:

* Glofitamab (a T-cell bispecific humanized monoclonal antibody)
* Obinutuzumab (a humanized glycoengineered type II anti-CD20 monoclonal antibody)
* Polatuzumab vedotin (an antibody-drug conjugate)
* Pirtobrutinib (a selective inhibitor of BTK)
* Atezolizumab (a humanized immunoglobulin monoclonal antibody)
* Tocilizumab (a recombinant, humanized, anti-human monoclonal antibody)

DETAILED DESCRIPTION:
This is an open-label, multicenter phase II study to evaluate the efficacy and safety of glofitamab as monotherapy and in combination with polatuzumab vedotin, pirtobrutinib, or atezolizumab for participants with Richter's Transformation (RT) that has transformed from chronic lymphocytic leukemia (CLL).

The U.S. Food and Drug Administration (FDA) has not approved glofitamab, obinutuzumab, polatuzumab vedotin, pirtobrutinib or atezolizumab for RT, but each drug has been approved for other uses.

Glofitamab has been approved by the FDA for certain people with diffuse large B-cell lymphoma (DLBCL), which is similar to Richter's Transformation. Glofitamab has been studied as a single therapy and in combination with polatuzumab vedotin and atezolizumab in people with DLBCL.

Polatuzumab vedotin is already an approved therapy for diffuse large B-cell lymphoma in combination with chemoimmunotherapy.

Pirtobrutinib is an approved therapy for chronic lymphocytic leukemia, small lymphocytic lymphoma, and mantle cell lymphoma.

Atezolizumab is an approved therapy for other cancers.

Obinutuzumab is an approved therapy for chronic lymphocytic leukemia.

Tocilizumab is approved for the treatment of an entity called cytokine release syndrome following another therapy called chimeric antigen receptor T-cell therapy; it will be used to treat cytokine release syndrome if a participant develops it in this study.

Study procedures include screening for eligibility, clinic visits for study treatment, blood and urine tests, Positron Emission Tomography (PET) or Computed Topography (CT) scans, bone marrow biopsies, echocardiograms, and electrocardiograms (ECGs).

Participants will receive study treatment for about 9 months and will be followed every 3-6 months for up to 10 years thereafter.

It is expected that about 70 people will take part in this research study.

Genentech, Inc./Loxo Oncology, Inc./Eli Lilly and Company are funding this research study by providing study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma as per IW-CLL 2018 criteria with biopsy proven transformation to diffuse large B-cell lymphoma (DLBCL), consistent with Richter's Transformation. The diagnostic sample must be reviewed by the treating institution. Tumor sample may be obtained by core needle or excisional surgical biopsy. A fresh biopsy is encouraged, but an archival sample is acceptable if the following provisions are met: 1) availability of a tumor-containing formalin-fixed, paraffin-embedded (FFPE) tissue block, 2) if the tumor containing FFPE tissue block cannot be provided in total, sections from this block should be provided. Biopsy can be obtained up to 3 months prior to first day of treatment.
* Cohort-specific eligibility criteria:

  * Glofitamab monotherapy cohort: Patients with either relapsed/refractory or previously untreated Richter's Transformation.
  * Glofitamab + polatuzumab vedotin cohort: Patients with previously untreated RT. After the first 10 patients are enrolled in this cohort irrespective of prior BTKi exposure status, the remainder of the patients enrolled to this cohort must have previously untreated RT and no prior BTK inhibitor. Patients cannot have prior polatuzumab vedotin exposure.
  * Glofitamab + pirtobrutinib cohort: Patients with previously untreated RT and prior BTK inhibitor exposure (with enrollment to begin only after the first 10 patients are accrued to the polatuzumab combination cohort). Patients cannot have prior pirtobrutinib exposure.
  * Glofitamab + atezolizumab cohort: Patients with relapsed/refractory RT. Patients are required to have received ≥ 1 prior line of therapy. Patients cannot have prior atezolizumab exposure.
* Age ≥18 years.
* ECOG performance status of 0-2 (Appendix A).
* For patients receiving glofitamab monotherapy, glofitamab in combination with polatuzumab vedotin, or glofitamab in combination with atezolizumab, participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count must be > 1.0 x10^9/L (growth factor allowed to achieve), unless patients have significant bone marrow involvement of their malignancy confirmed on biopsy.
  * Platelets must be > 30 x10^9/L, independent of transfusion within 7 days of screening, unless patients have bone marrow involvement of their malignancy confirmed on biopsy
  * Creatinine < 2.0 x ULN (upper limit of normal) or estimated CrCl > 50 ml/min
  * Total bilirubin < 1.5 X ULN
  * Subjects with Gilbert's Syndrome or resolving autoimmune hemolytic anemia may have a bilirubin up to 3.0 X ULN
  * AST/ALT < 3.0 X ULN, unless documented liver involvement by lymphoma
* For patients receiving glofitamab in combination with pirtobrutinib, participants must meet the following:

  * Absolute neutrophil count must be > 1.0 x109/L (growth factor >7 days prior allowed to achieve), unless patients have significant bone marrow involvement of their malignancy confirmed on biopsy.
  * Hemoglobin > 8 g/dL, independent of transfusion within 7 days of screening, unless patients have bone marrow involvement of their malignancy confirmed on biopsy
  * Platelets must be > 50 x109/L, independent of transfusion within 7 days of screening
  * Estimated CrCl > 50 ml/min according to Cockcroft/Gault formula
  * AST/ALT < 3.0 X ULN, or < 5.0 X ULN with documented liver involvement by lymphoma
  * Total bilirubin < 1.5 X ULN or < 3.0 x ULN with documented liver involvement by lymphoma and/or Gilbert's Disease
  * Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x ULN.
  * The patient is able to take oral medications
* Patients who have undergone prior allogeneic transplantation are potentially eligible if their transplant day 0 is > 6 months from their first dose of treatment and as follows:

  * For patients receiving glofitamab monotherapy or glofitamab in combination with polatuzumab vedotin, all of the following must additionally be true:

    * No current or prior Grade 3/4 graft versus host disease (GVHD)
    * Stable off of immunosuppression for at least 2 months prior to receiving their first dose of treatment on study
  * For patients receiving glofitamab in combination with pirtobrutinib, all of the following must additionally be true:

    * No active/current GVHD
    * No prior history of Grade 3/4 GVHD
    * Stable off of immunosuppression for at least 2 months prior to receiving their first dose of treatment on study
  * For patients receiving atezolizumab, no prior allogeneic hematopoietic cell transplantation is allowed.
* Willingness to remain abstinent (refrain from heterosexual intercourse) or to use effective contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least the following durations listed below:

  * Female patients: at least 18 months after pre-treatment with obinutuzumab, or 2 months after the last dose of glofitamab, or 5 months after the last dose of atezolizumab, or 9 months after the last dose of polatuzumab vedotin, 3 months after the last dose of tocilizumab (if applicable), or 1 month after the last dose of pirtobrutinib, whichever whichever is longest.
  * Male patients: at least 3 months after pre-treatment with obinutuzumab, or 2 months after the last dose of glofitamab, or 5 months after the last dose of polatuzumab vedotin, or 2 months after the last dose of tocilizumab (if applicable), whichever is longest.
  * Examples of highly effective contraceptive methods with a failure rate of <1% per year include: Tubal ligation, male sterilization, hormonal implants, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide.
* For female patients, willingness to refrain from donating ova during the same periods described in section 3.1.6 for female patients. For male patients, willingness to refrain from donating sperm during the same periods described in section 3.1.6 for male patients.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Patients with the Hodgkin variant transformation of CLL will be excluded.
* No prior anti-CD20 bispecific antibody is allowed. No prior, polatuzumab vedotin is allowed for patients in the polatuzumab vedotin-containing combination arm. No prior, or atezolizumab therapy is allowed for patients in the atezolizumab-containing combination arm. No prior pirtobrutinib is allowed for patients in the pirtobrutinib-containing arm.
* Subject has received any of the following within 14 days or 5 drug half-lives (whichever is shortest) prior to the first dose of treatment: investigational agents, targeted therapies, e.g. tyrosine kinase inhibitors, systemic immunotherapeutic/immunostimulating agents, including, but not limited to, CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, radio-immunoconjugates, antibody-drug conjugates (patients in the pirtobrutinib combination arm may not have received an antibody-drug conjugate within 28 days prior to the first dose of study treatment), immune/cytokines and monoclonal antibodies. Patients who are currently receiving treatment with a Bruton's tyrosine kinase inhibitor may continue this agent until the day prior to starting treatment, to reduce the risk of tumor flare on treatment cessation.
* Prior treatment with CAR T-cell therapy within 30 days before first study treatment administration.
* Subject has not recovered to less than Grade 1 clinically significant adverse effect(s)/toxicity from prior anti-cancer therapy including immunotherapy, with the exception of alopecia, endocrinopathy managed with replacement therapy, and stable vitiligo.
* Patients with bulky cervical adenopathy that is compressing the upper airway and could result in significant further airway compression during a tumor flare event.
* History of other malignancies, except:

  * CLL/SLL
  * Malignancy treated with curative intent and with no known active disease present before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Low-risk prostate cancer on active surveillance
* For patients receiving polatuzumab vedotin: Current > Grade 1 peripheral neuropathy.
* Any history of immune-related ≥ Grade 3 AE with the exception of endocrinopathy managed with replacement therapy.
* Patient with history of confirmed progressive multifocal leukoencephalopathy (PML).
* Current or past history of central nervous system (CNS) disease involvement or history of leptomeningeal disease.
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease (Note: patients with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits, as judged by the investigator, are permitted).
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
* Prior solid organ transplantation.
* History of known or suspected hemophagocytic lymphohistiocytosis (HLH).
* Active or history of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  * Patients with a remote history of, or well controlled, autoimmune disease may be eligible to enroll after consultation with the study PI.
  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone and patients with controlled Type 1 diabetes mellitus who are on an insulin regimen can be included.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided that the disease is well controlled (Rash <10% of BSA, and no acute exacerbations requiring methotrexate, retinoids, biologics, or high potency oral corticosteroids) at baseline and requires only low-potency topical corticosteroids.
  * For patients enrolling to the pirtobrutinib combination arm, patients with the following should be discussed with the Sponsor-Investigator prior to enrollment: active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
* Patients who require systemic immunosuppressive therapy for an ongoing medical condition will be excluded with the exception of corticosteroid use for disease-related symptom control. Treatment for autoimmune disease with systemic immunosuppressive medications including, but not limited to, prednisone, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents are not allowed within 2 weeks prior to Day 1 of Cycle 1.

  * Note the following are permitted: use of inhaled corticosteroids, use of mineralocorticoids for management of orthostatic hypotension.
  * Corticosteroids for lymphoma symptom control is allowed provided patients are on a stable dose as per discretion of the treating investigator and in discussion with the Sponsor-Investigator.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy unless in consultation with an allergy specialist they are deemed eligible for retreatment with desensitization.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
* History of Human Immunodeficiency Virus (HIV):

  * For patients receiving glofitamab in combination with pirtobrutinib, patients who have tested positive for HIV are excluded due to risk of opportunistic infections with both HIV and BTK inhibitors. For patients with unknown HIV status, HIV testing will be performed at screening and result must be negative for enrollment.
  * For patients in all other cohorts, only those without controlled disease (controlled disease defined as CD4 count greater than or equal to 200 per microliter, undetectable viral load, and stable anti-retroviral therapy) will be excluded.
* History of Human T-Cell Leukemia Virus 1 (HTLV-1) infection.
* Known active cytomegalovirus (CMV) infection.
* Clinically significant liver disease, including cirrhosis and active viral or non-viral hepatitis. Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative viral load (by PCR testing), be willing to undergo regular testing, and be able to be treated with a prophylactic agent (e.g. entecavir). Patients with hepatitis C seropositivity are eligible only if they have a negative viral load (by PCR testing).
* Patients with a known active infection or any major episode of infection requiring hospitalization or treatment with IV antimicrobial within 4 weeks prior to first study drug. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation), antivirals, or antifungals may participate.
* Patients should not have received immunization with live vaccines within 28 days prior to start of study treatment. In addition, patients must not receive live, attenuated vaccines (e.g., FluMist®) while receiving study treatment or after the last dose until B-cell recovery to the normal ranges. Inactivated influenza vaccination is permitted during influenza season.
* Patients with any one of the following currently or in the previous 6 months will be excluded: myocardial infarction, congenital long QT syndrome, torsade de pointes, unstable angina, or coronary/peripheral artery bypass graft.
* Patients with New York Heart Association Class III or IV heart failure or with Objective Assessment Class C or D cardiac disease.
* For patients receiving pirtobrutinib:

  * Significant cardiovascular disease defined as:

    * unstable angina or acute coronary syndrome within the past 2 months prior to randomization
    * history of myocardial infarction within 3 months prior to randomization or
    * documented LVEF by any method of ≤ 40% in the 12 months prior to randomization
  * Uncontrolled or symptomatic arrhythmias

    * Note: patients with atrial fibrillation are allowed as long as they are adequately rate-controlled.)
    * Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
  * Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33).

    * Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
    * Correction for underlying bundle branch block (BBB) allowed.
  * Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug.
  * Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
  * Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.
  * Have a known hypersensitivity to any of the excipients of Pirtobrutinib or to any intended study medications.
  * Patients who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor. Note: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
  * History of bleeding disorders (e.g. von Willebrand's disease, hemophilia).
  * History of stroke or intracranial hemorrhage within 6 months of starting study therapy.
* Inability to comply with protocol mandated hospitalizations and restrictions.
* Patients who are pregnant, breast-feeding, or intending to become pregnant during the study.
* Any other diseases, metabolic dysfunction, physical examination finding, mental status or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2033-01-15 (Estimated)

PRIMARY OUTCOMES:
Best Complete Response (CR) Rate | Disease evaluation will be performed at 12, 24 and 36 weeks
  Best Complete Response (CR) rate is defined as the proportion of participants achieving CR at any of the 3 timepoints (after 4, 8 and 12 cycles). CR is defined per Lugano 2014 criteria.

SECONDARY OUTCOMES:
Best Overall Response Rate (ORR) | Disease evaluation will be performed at 12, 24 and 36 weeks
  Best Overall response rate (ORR) is defined as the proportion of participants achieving complete response (CR) or partial response (PR) at any of the 3 timepoints (after 4, 8 and 12 cycles). CR and PR are defined per Lugano 2014 criteria.
Best Partial Response (PR) Rate | Disease evaluation will be performed at 12, 24 and 36 weeks
  Best Partial response (PR) rate is defined as the proportion of participants achieving partial response at any of the 3 timepoints (after 4, 8, 12 cycles). PR is defined per Lugano 2014 criteria.
Overall Response Rate at 36 weeks | 36 weeks
  Overall response rate (ORR) at 36 weeks is defined as the proportion of participants who achieve complete response (CR) or partial response (PR) at the time of disease evaluation at 12 cycles (36 weeks). CR and PR are defined per Lugano 2014 criteria.
Partial Response (PR) Rate at 36 weeks | 36 weeks
  Partial Response (PR) rate at 36 weeks is defined as the proportion of participants achieving PR at the time of disease evaluation at 12 cycles (36 weeks). PR defined per Lugano 2014 criteria.
Complete Response (CR) Rate at 36 weeks | 36 weeks
  Complete Response (CR) rate at 36 weeks is defined as the proportion of participants achieving CR at the time of disease evaluation at 12 cycles (36 weeks). CR defined per Lugano 2014 criteria.
Duration of Response (DOR) | Disease evaluation will be performed every 3 months, up to 2 years.
  Duration of Response (DOR) is defined as the time from date of first documented confirmed objective response (CR + PR) to date of first documented progressive disease (PD) per Lugano 2014 criteria.
Duration of Complete Response (DOCR) | In long-term follow-up, participants were assessed every 6 months, up to 2 years
  Duration of complete response (DOCR) is defined as the time from date of first documented complete response to date of first documented progressive disease (PD) per Lugano 2014 criteria.
Progression Free Survival (PFS) at 2 years | Participants will be followed up to 2 years.
  PFS at 2 years is the percent probability estimate at 2 years based on the Kaplan-Meier method. PFS will be calculated as the time from start of treatment to the date of progressive disease (PD, defined per Lugano 2014 criteria), death, or last follow-up. Participants alive and progression-free at time of last follow-up will be censored.
Median Progression Free Survival (PFS) | Participants will be followed up to 2 years.
  PFS will be calculated as the time from start of treatment to the date of progressive disease (PD, defined per Lugano 2014 criteria), death, or last follow-up. Participants alive and progression-free at time of last follow-up will be censored.
Overall Survival (OS) at 2 years | Participants will be followed up to 2 years.
  OS at 2 years is the percent probability at 2 years based on Kaplan-Meier methodology. OS will be calculated as the time from the start of treatment to the date of death, or last follow-up. Participants alive at time of last follow-up will be censored.
Median Overall Survival | Participants will be followed up to 10 years.
  OS will be calculated as the time from the start of treatment to the date of death, or last follow-up. Participants alive at time of last follow-up will be censored.
Minimal Residual Disease (MRD) Negativity | MRD testing will be performed every 3 months, up to 2 years, then every 6 months, up to 3 years (5 years in total)
  MRD negativity is defined as the proportion of participants that achieve MRD negative, where it measured by multiparametric flow cytometry (Mayo Clinic Laboratories) or the clonoSEQ assay (Adaptive).
Rate and severity of Cytokine Release Syndrome (CRS), immune effector cell-associated Neurotoxicity Syndrome (ICANS), and Hemophagocytic Lymphohistiocyotis (HLH) | Adverse events will be collected at each study visit plus 30 days post treatment end, up to 10 months.
  CRS, ICANS, and HLH rates and severity will be summarized based on American Society of Transplantation and Cellular Therapy (ASTCT) Consensus grading.
Tocilizumab Usage Rate | Within the first year on study
  Tocilizumab usage rate is defined as the proportion of participants requiring tocilizumab usage of management of CRS.
Median Tocilizumab Usage | Within the first year on study
  Median tocilizumab usage is defined as median number of doses of tocilizumab administered per participant
Grade 3-5 Adverse Events Rate | Adverse events will be collected at each study visit plus 30 days post treatment end
  Grade 3-5 AE rate is defined as the proportion of patients who experienced grade 3-5 adverse event based on the Common Toxicity Criteria for Adverse Events version 5.0 as reported on case report form.
Treatment-related Adverse Events Rate | Adverse events will be collected at each study visit plus 30 days post treatment end
  Treatment-related adverse event rate is defined as the proportion of participants who experienced treatment-related adverse event based on the Common Toxicity Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ryan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu